CLINICAL TRIAL: NCT05832788
Title: Occupational Hazards and Associated Health Effects Among Workers in Main Assiut University Printing Press
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fatma EL Zahraa Mohamed Hussein Ahmed (Other)
Responsible Party: Sponsor-Investigator, Fatma EL Zahraa Mohamed Hussein Ahmed, demonstrator, Assiut University
Organization: Assiut University (Other)
Other Study IDs: printing hazards
Record Dates: First submitted 2023-03-29; First posted 2023-04-27 (Actual); Last update posted 2023-04-27 (Actual); Status verified 2023-04

CONDITIONS: Printing Hazards

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Occupational Hazards and Associated Health Effects among Workers in Main Assiut University Printing Press

DETAILED DESCRIPTION:
Printing in its simplest forms has existed for thousands of years, in the form of signet rings, royal seals and punches used by gold and silver-smiths.

Each printing process is divided into 3 major steps: prepress, press, and post-press. Prepress operations include the composition, typesetting, graphic arts photography, assembly of images and preparation of image carrier. Press includes the actual printing operation. Post-press involves the assembly of printed materials, binding and finishing operations.

Workers in printing press are exposed to, chemical, physical, ergonomic, and psychological hazards.

Chemical hazards are the most serious one. due to exposure to lot of chemical substances such as organic solvents, inks, adhesives, organic and inorganic pigments, The most important chemical substances used are Volatile Organic compounds, and inks.

Exposure to these chemicals occurs through both inhalation and dermal contact, The Acute symptoms include dizziness, drowsiness, eye irritation,.etc. Long-term health effects may include damage of internal organs as liver, kidneys and lungs, brain, reproductive system, bladder etc.

Dermatitis is a common health effect among printing workers due to exposure to chemicals.

One of the intended components of inks, solvents, and cleaning agents form is Benzene, long term exposure to benzene cause blood disorders. It specifically affects bone marrow, thus leading to decrease in the erythrocytes and leukocytes production resulting in anemia, myeloid leukemia, thrombocytopenia.

Noise is health hazard to which those workers are exposed, it occurs during printing, binding, folding.

Ergonomic hazards are hazards among those workers in the form of serious accidents and musculoskeletal disorders.

ELIGIBILITY:
Inclusion Criteria:

* 1. Workers with more than one year work duration.
* 2. both sexes, males and females.

Exclusion Criteria:

- 1. Workers who have any blood health problems as blood cells disorders and bleeding disorders before they started working.

2. Pre-employment liver diseases and kidney diseases among those workers. 3. Workers with less than one year work duration.

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Main Assiut University Printing Press workers.
Sampling Method: Probability Sample
Enrollment: 83 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-10-01 (Estimated)

PRIMARY OUTCOMES:
• Describe the occupational hazards and associated negative health effects of these hazards among workers at Main Assiut University Printing Press. | 3 years
  • Laboratory investigations and questionnaire will be used to assess this measure

SECONDARY OUTCOMES:
• Identify associated risk factors to these effects among the study workers. | 3 years
  • questionnaire will be used to assess this measure